CLINICAL TRIAL: NCT05668260
Title: Internal Biodegradable Stent Versus Non-Stent in Patients at High-Risk of Developing Fistula After Pancreatoduodenectomy (BioSteP): a Randomized Controlled Study
Brief Title: Internal Biodegradable Stent Versus Non-Stent in Patients at High-Risk of Developing Fistula After Pancreatoduodenectomy
Acronym: BioSteP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: amg International (Unknown)
Responsible Party: Principal Investigator, Stefano Partelli, Professor, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BioSteP
Record Dates: First submitted 2022-12-12; First posted 2022-12-29 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pancreatoduodenectomy; Clinically Relevant Postoperative Pancreatic Fistula; Internal Biodegradable Pancreatic Stent
Keywords: Pancreatic surgery; Pancreatoduodenectomy; CR-POPF; Post operative complications; ARCHIMEDES™

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biodegradable Stent (Experimental): An internal biodegradable pancreatic stent (ArchimedesTM) will be placed at the level of the pancreatic anastomosis in patients undergoing pancreatoduodenectomy.
  Interventions: Device: Biodegradable Stent
- Non Stent (No Intervention): No stent will be placed at the level of the pancreatic anastomosis in patients undergoing pancreatoduodenectomy.

INTERVENTIONS:
Device: Biodegradable Stent — A trans-anastomotic biodegradable internal stent (ARCHIMEDES™) will be placed between the main pancreatic duct (MPD) and the enterotomy in the jejunum just after the completion of the posterior suture of duct-to-mucosa. The biodegradable stent will then be shaped according to the angle of the jejunal loop in order to minimise the risk of displacement. The adequate length of the stent will be chosen according to the length of the jejunal loop.
  Arms: Biodegradable Stent

SUMMARY:
The aim of this randomized controlled study is to compare the efficacy of biodegradable internal pancreatic stenting versus no stenting in patients undergoing pancreatoduodenectomy (PD), focusing on a possible superiority association of the device in preventing clinically relevant postoperative pancreatic fistula (CR-POPF).

Patients undergoing PD will be randomized into two arms:

* arm 1: a biodegradable internal pancreatic stent will be placed at the level of the pancreatic anastomosis
* arm 2: no pancreatic stent will be placed at the level of the pancreatic anastomosis

The rate of occurrence of CR-POPF will be compared between the two arms.

DETAILED DESCRIPTION:
Clinically relevant postoperative pancreatic fistula (CR-POPF) represents the most common complication that can occur after pancreatoduodenectomy (PD). CR-POPF is the main cause of morbidity after PD, being associated with a risk of mortality up to 60%. The placement of external or internal pancreatic stents after PD have been investigated as possible strategies for preventing the development of CR-POPF. However, device displacement has been reported as a common cause of pancreatic stents malfunction. Recently, a novel biodegradable pancreatic stent (ARCHIMEDES™) has been introduced. The device has been specifically designed to reduce the risk of displacement, thus offering a new valuable tool to decrease the rate of CR-POPF after PD.

In this randomised, controlled, single-center trial, researchers investigate the possible efficacy of biodegradable internal pancreatic stenting of pancreatic anastomosis in patient undergoing PD versus no stenting, focusing on a possible superiority association for preventing CR-POPF.

Participants will be randomised into two arms (Biodegradable stent vs non-stent) based on their intra-operative risk of developing POPF according to the Fistula Risk Score (FRS). The rate of CR-POPF will be compared between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Patients who undergo pancreatoduodenectomy (PD)
* Informed Consent

Exclusion Criteria:

* Previous distal pancreatectomy
* Patients with intra-operative negligible, intermediate or moderate risk of POPF (fistula risk score < 7)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Clinically Relevant Postoperative Pancreatic Fistula (CR-POPF) | from three days after surgery until 3 months after surgery
  The primary objective of the study is to compare the rate of CR-POPF after PD with duct-to-mucosa pancreatico-jejunostomy (PJ) using biodegradable pancreatic internal stent vs no stent.

SECONDARY OUTCOMES:
Clinically Relevant Postoperative Pancreatic Fistula (CR-POPF) severity | from three days after surgery until 3 months after surgery
  The difference between the two treatment arms in terms of severity of CR-POPF will be assessed. CR-POPF will be classified according to the ISGPS definition into two groups: grade B and grade C. Grade B will be further sub-classified in three categories according to Maggino et al.: grade B1, grade B2, grade B3.
Postoperative Morbidity | from the date of surgery, up to 3 months
  The difference between the two treatment arms in terms of rate of overall postoperative morbidity as defined by Dindo et al. will be assessed. Additionally the Comprehensive Complication Index will be calculated. Post-pancreatectomy hemorrhage (PPH) and delayed gastric emptying (DGE) will be defined according to ISGPS definitions.
Length of Hospital Stay (LOS) | from the date of surgery until the date of hospital discharge, assessed up to 3 months
  The difference between the two treatment arms in terms of median LOS will be assessed. Median LOS will be defined by subtracting the date of surgery from the date when the enrolled patients are discharged from the hospital.
Time to Functional Recovery (TFR) | from the date of surgery until the date of functional recovery, assessed up to 3 months
  The difference between the two treatment arms in terms of time to functional recovery (TFR) will be assessed. TFR will be defined by subtracting the date of surgery from the date when participants achieve standardized criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilise and self-care and no evidence of untreated medical problems).
Quality of Life (QoL) | from the day before surgery until 3 months after surgery
  The difference between the two treatment arms in terms of QoL will be assessed. QoL will be measured in several ways. First, self-reported activity status will be measured using the Duke Activity Status Index (Duke Index, DASI)., a brief questionnaire designed to assess physical function and predict exercise capacity (peak oxygen uptake). Second, generic health related QoL will be measured using the Patient Reported Outcome Measure Information System (PROMIS)-29+2 Profile v2.1 (PROPr), a questionnaire designed to measure self-reported physical, mental and social health and wellbeing.
Cost-effectiveness | from the date of surgery, up to 3 months
  The difference between the two treatment arms in terms of cost-effectiveness will be assessed. Cost-effectiveness will be estimated by the ration of differences in costs to differences in quality adjusted life years (QALYs) between the two groups of the study. QALYs will be calculated using the preference scores obtained from PROMIS-29+2. To calculate QALYs, the preference scores at 90 days after surgery will be multiplied by 0.25 (which represents 1/4 of the year). Cost of care will be estimated considering resources consumed during hospital stay and use of healthcare resources after hospital discharge.
Stent displacement | 10 days after surgery
  The rate of biodegradable rate displacement as detected by postoperative contrast-enhanced computed tomography (CE-CT) performed by 10 days after surgery. A displacement will be defined by the absence of visible trans-anastomotic stent or by its complete dislocation in the jejunum/ileum or colon.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Marchegiani G, Andrianello S, Salvia R, Bassi C. Current Definition of and Controversial Issues Regarding Postoperative Pancreatic Fistulas. Gut Liver. 2019 Mar 15;13(2):149-153. doi: 10.5009/gnl18229. PMID 30419630
- [Background] Partelli S, Andreasi V, Schiavo Lena M, Rancoita PMV, Mazza M, Mele S, Guarneri G, Pecorelli N, Crippa S, Tamburrino D, Doglioni C, Falconi M. The role of acinar content at pancreatic resection margin in the development of postoperative pancreatic fistula and acute pancreatitis after pancreaticoduodenectomy. Surgery. 2021 Oct;170(4):1215-1222. doi: 10.1016/j.surg.2021.03.047. Epub 2021 Apr 28. PMID 33933282
- [Background] Smits FJ, Molenaar IQ, Besselink MG, Borel Rinkes IHM, van Eijck CHJ, Busch OR, van Santvoort HC; Dutch Pancreatic Cancer Group. Early recognition of clinically relevant postoperative pancreatic fistula: a systematic review. HPB (Oxford). 2020 Jan;22(1):1-11. doi: 10.1016/j.hpb.2019.07.005. Epub 2019 Aug 21. PMID 31445782
- [Background] Shrikhande SV, Sivasanker M, Vollmer CM, Friess H, Besselink MG, Fingerhut A, Yeo CJ, Fernandez-delCastillo C, Dervenis C, Halloran C, Gouma DJ, Radenkovic D, Asbun HJ, Neoptolemos JP, Izbicki JR, Lillemoe KD, Conlon KC, Fernandez-Cruz L, Montorsi M, Bockhorn M, Adham M, Charnley R, Carter R, Hackert T, Hartwig W, Miao Y, Sarr M, Bassi C, Buchler MW; International Study Group of Pancreatic Surgery (ISGPS). Pancreatic anastomosis after pancreatoduodenectomy: A position statement by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2017 May;161(5):1221-1234. doi: 10.1016/j.surg.2016.11.021. Epub 2016 Dec 24. PMID 28027816
- [Background] Nahm CB, Connor SJ, Samra JS, Mittal A. Postoperative pancreatic fistula: a review of traditional and emerging concepts. Clin Exp Gastroenterol. 2018 Mar 15;11:105-118. doi: 10.2147/CEG.S120217. eCollection 2018. PMID 29588609
- [Background] Xiong JJ, Altaf K, Mukherjee R, Huang W, Hu WM, Li A, Ke NW, Liu XB. Systematic review and meta-analysis of outcomes after intraoperative pancreatic duct stent placement during pancreaticoduodenectomy. Br J Surg. 2012 Aug;99(8):1050-61. doi: 10.1002/bjs.8788. Epub 2012 May 24. PMID 22622664
- [Background] Dong Z, Xu J, Wang Z, Petrov MS. Stents for the prevention of pancreatic fistula following pancreaticoduodenectomy. Cochrane Database Syst Rev. 2016 May 6;2016(5):CD008914. doi: 10.1002/14651858.CD008914.pub3. PMID 27153248
- [Background] Pessaux P, Sauvanet A, Mariette C, Paye F, Muscari F, Cunha AS, Sastre B, Arnaud JP; Federation de Recherche en Chirurgie (French). External pancreatic duct stent decreases pancreatic fistula rate after pancreaticoduodenectomy: prospective multicenter randomized trial. Ann Surg. 2011 May;253(5):879-85. doi: 10.1097/SLA.0b013e31821219af. PMID 21368658
- [Background] Andrianello S, Marchegiani G, Malleo G, Masini G, Balduzzi A, Paiella S, Esposito A, Landoni L, Casetti L, Tuveri M, Salvia R, Bassi C. Pancreaticojejunostomy With Externalized Stent vs Pancreaticogastrostomy With Externalized Stent for Patients With High-Risk Pancreatic Anastomosis: A Single-Center, Phase 3, Randomized Clinical Trial. JAMA Surg. 2020 Apr 1;155(4):313-321. doi: 10.1001/jamasurg.2019.6035. PMID 32101272
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Braga M, Pecorelli N, Ariotti R, Capretti G, Greco M, Balzano G, Castoldi R, Beretta L. Enhanced recovery after surgery pathway in patients undergoing pancreaticoduodenectomy. World J Surg. 2014 Nov;38(11):2960-6. doi: 10.1007/s00268-014-2653-5. PMID 24870390
- [Background] Maggino L, Malleo G, Bassi C, Allegrini V, McMillan MT, Borin A, Chen B, Drebin JA, Ecker BL, Fraker DL, Lee MK, Paiella S, Roses RE, Salvia R, Vollmer CM Jr. Decoding Grade B Pancreatic Fistula: A Clinical and Economical Analysis and Subclassification Proposal. Ann Surg. 2019 Jun;269(6):1146-1153. doi: 10.1097/SLA.0000000000002673. PMID 31082914
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Background] Alonso J, Permanyer-Miralda G, Cascant P, Brotons C, Prieto L, Soler-Soler J. Measuring functional status of chronic coronary patients. Reliability, validity and responsiveness to clinical change of the reduced version of the Duke Activity Status Index (DASI). Eur Heart J. 1997 Mar;18(3):414-9. doi: 10.1093/oxfordjournals.eurheartj.a015260. PMID 9076377